CLINICAL TRIAL: NCT06146764
Title: Contrast-enhanced Ultrasound Improves the Diagnostic Performance of Sonographic Risk Stratification System of Thyroid Carcinoma: Comparison Between Integrated Scoring Method and Up-and-down Scoring Method
Brief Title: CEUS Improves the Diagnostic Performance of SRSS of Thyroid Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jingliang Ruan, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-1024-01
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Nodule; Thyroid Carcinoma
Keywords: Thyroid Nodule; Contrast Media; Gray-scale Ultrasound; Diagnosis; Biopsy
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced Ultrasound — Integrated scoring method and up-and-down scoring method

SUMMARY:
Contrast-enhanced ultrasound (CEUS) can sensitively show the blood perfusion characteristics of thyroid nodules, which is a useful supplement to gray-scale ultrasound. However, there is no standard combined diagnostic method of gray-scale ultrasound and CEUS. Therefore, the aim of this study was to compare the diagnostic performance of the integrated scoring method and the up-and-down scoring method. This study was a multicenter retrospective clinical study and followed the Standards for Reporting of Diagnostic Accuracy Studies (version 2015). Inclusion criteria: 1) participants with at least one thyroid nodule larger than 5 mm confirmed by conventional ultrasound; 2) participants underwent gray-scale ultrasound, contrast-enhanced ultrasound and fine needle aspiration biopsy of the thyroid nodule successively; 3) participants have a final diagnosis of benign or malignant. Exclusion criteria included: 1) participants with cytologic findings of Bethesda I, III, or IV without definitive benign or malignant pathologic findings; 2) participants with a history of thyroid fine needle aspiration, ablation or surgery; 3) participants with low quality ultrasound images (e.g., severe artifacts or low image resolution). According to the American College of Radiology Thyroid Imaging Reporting and Data System, only one thyroid nodule with the highest point was included in each participant. A total of 600 participants from January 2018 to December 2022 were consecutively included in Sun Yat-sen Memorial Hospital of Sun Yat-sen University to form a training set (average age 48 years; Range 24-81 years old). A total of 200 subjects with thyroid nodules from January 2022 to December 2022 were consecutively included to form an external validation set in Houjie Hospital of Dongguan City, Guangdong Province (mean age 46 years; Range 30-74 years). The malignant risk of enrolled thyroid nodules and the necessity of biopsy were evaluated by integrated scoring method and up-and-down scoring method, respectively. The diagnostic performance and unnecessary biopsy rate of the above two methods were calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Participants with thyroid nodules with a solid component ≥5 mm confirmed by conventional ultrasound;
* Participants who underwent conventional ultrasound, contrast-enhanced ultrasound, and fine-needle aspiration biopsy;
* Participants with a final benign or malignant pathological results.

Exclusion Criteria:

* Participants with cytopathology of Bethesda I, III, or IV and without final benign or malignant pathology；
* Participants with a history of thyroid ablation or surgery;
* Participants with low-quality ultrasound images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included patients at Sun Yat-sen Memorial Hospital (the internal validation set) and Houjie Hospital of Dongguan(the external validation set) at the same eligibility criteria described above from January 2021 to December 2022.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | First week after primary completion date
  Sensitivity, specificity, positive predictive value, negative predictive value, area under the curve
Unnecessary biopsy rate | First week after primary completion date
  The unnecessary biopsy rate was defined as a percentage of the number of benign nodules among biopsy-indicated nodules in the total nodules.

CONTACTS AND LOCATIONS:
Overall Officials: Jingliang Ruan, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Baoming Luo, Professor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data generated or analyzed during the study are available from the principal investigator by request.
Supporting Information: Study Protocol
Time Frame: The first week after the publication of the research papers.
Access Criteria: Data generated or analyzed during the study are available from the principal investigator by request.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Pizzato M, Li M, Vignat J, Laversanne M, Singh D, La Vecchia C, Vaccarella S. The epidemiological landscape of thyroid cancer worldwide: GLOBOCAN estimates for incidence and mortality rates in 2020. Lancet Diabetes Endocrinol. 2022 Apr;10(4):264-272. doi: 10.1016/S2213-8587(22)00035-3. Epub 2022 Mar 7. PMID 35271818
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Zhou J, Yin L, Wei X, Zhang S, Song Y, Luo B, Li J, Qian L, Cui L, Chen W, Wen C, Peng Y, Chen Q, Lu M, Chen M, Wu R, Zhou W, Xue E, Li Y, Yang L, Mi C, Zhang R, Wu G, Du G, Huang D, Zhan W; Superficial Organ and Vascular Ultrasound Group of the Society of Ultrasound in Medicine of the Chinese Medical Association; Chinese Artificial Intelligence Alliance for Thyroid and Breast Ultrasound. 2020 Chinese guidelines for ultrasound malignancy risk stratification of thyroid nodules: the C-TIRADS. Endocrine. 2020 Nov;70(2):256-279. doi: 10.1007/s12020-020-02441-y. Epub 2020 Aug 21. PMID 32827126
- [Background] Tessler FN, Middleton WD, Grant EG, Hoang JK, Berland LL, Teefey SA, Cronan JJ, Beland MD, Desser TS, Frates MC, Hammers LW, Hamper UM, Langer JE, Reading CC, Scoutt LM, Stavros AT. ACR Thyroid Imaging, Reporting and Data System (TI-RADS): White Paper of the ACR TI-RADS Committee. J Am Coll Radiol. 2017 May;14(5):587-595. doi: 10.1016/j.jacr.2017.01.046. Epub 2017 Apr 2. PMID 28372962
- [Background] Russ G, Bonnema SJ, Erdogan MF, Durante C, Ngu R, Leenhardt L. European Thyroid Association Guidelines for Ultrasound Malignancy Risk Stratification of Thyroid Nodules in Adults: The EU-TIRADS. Eur Thyroid J. 2017 Sep;6(5):225-237. doi: 10.1159/000478927. Epub 2017 Aug 8. PMID 29167761
- [Background] Shin JH, Baek JH, Chung J, Ha EJ, Kim JH, Lee YH, Lim HK, Moon WJ, Na DG, Park JS, Choi YJ, Hahn SY, Jeon SJ, Jung SL, Kim DW, Kim EK, Kwak JY, Lee CY, Lee HJ, Lee JH, Lee JH, Lee KH, Park SW, Sung JY; Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. Ultrasonography Diagnosis and Imaging-Based Management of Thyroid Nodules: Revised Korean Society of Thyroid Radiology Consensus Statement and Recommendations. Korean J Radiol. 2016 May-Jun;17(3):370-95. doi: 10.3348/kjr.2016.17.3.370. Epub 2016 Apr 14. PMID 27134526
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Perros P, Boelaert K, Colley S, Evans C, Evans RM, Gerrard Ba G, Gilbert J, Harrison B, Johnson SJ, Giles TE, Moss L, Lewington V, Newbold K, Taylor J, Thakker RV, Watkinson J, Williams GR; British Thyroid Association. Guidelines for the management of thyroid cancer. Clin Endocrinol (Oxf). 2014 Jul;81 Suppl 1:1-122. doi: 10.1111/cen.12515. No abstract available. PMID 24989897
- [Background] Wemeau JL, Sadoul JL, d'Herbomez M, Monpeyssen H, Tramalloni J, Leteurtre E, Borson-Chazot F, Caron P, Carnaille B, Leger J, Do C, Klein M, Raingeard I, Desailloud R, Leenhardt L. Guidelines of the French society of endocrinology for the management of thyroid nodules. Ann Endocrinol (Paris). 2011 Sep;72(4):251-281. doi: 10.1016/j.ando.2011.05.003. Epub 2011 Jul 22. PMID 21782154
- [Background] Frates MC, Benson CB, Charboneau JW, Cibas ES, Clark OH, Coleman BG, Cronan JJ, Doubilet PM, Evans DB, Goellner JR, Hay ID, Hertzberg BS, Intenzo CM, Jeffrey RB, Langer JE, Larsen PR, Mandel SJ, Middleton WD, Reading CC, Sherman SI, Tessler FN; Society of Radiologists in Ultrasound. Management of thyroid nodules detected at US: Society of Radiologists in Ultrasound consensus conference statement. Radiology. 2005 Dec;237(3):794-800. doi: 10.1148/radiol.2373050220. PMID 16304103
- [Background] Middleton WD, Teefey SA, Reading CC, Langer JE, Beland MD, Szabunio MM, Desser TS. Comparison of Performance Characteristics of American College of Radiology TI-RADS, Korean Society of Thyroid Radiology TIRADS, and American Thyroid Association Guidelines. AJR Am J Roentgenol. 2018 May;210(5):1148-1154. doi: 10.2214/AJR.17.18822. Epub 2018 Apr 9. PMID 29629797
- [Background] Hoang JK, Middleton WD, Farjat AE, Langer JE, Reading CC, Teefey SA, Abinanti N, Boschini FJ, Bronner AJ, Dahiya N, Hertzberg BS, Newman JR, Scanga D, Vogler RC, Tessler FN. Reduction in Thyroid Nodule Biopsies and Improved Accuracy with American College of Radiology Thyroid Imaging Reporting and Data System. Radiology. 2018 Apr;287(1):185-193. doi: 10.1148/radiol.2018172572. Epub 2018 Mar 2. PMID 29498593
- [Background] Radzina M, Ratniece M, Putrins DS, Saule L, Cantisani V. Performance of Contrast-Enhanced Ultrasound in Thyroid Nodules: Review of Current State and Future Perspectives. Cancers (Basel). 2021 Oct 30;13(21):5469. doi: 10.3390/cancers13215469. PMID 34771632
- [Background] Ruan J, Xu X, Cai Y, Zeng H, Luo M, Zhang W, Liu R, Lin P, Xu Y, Ye Q, Ou B, Luo B. A Practical CEUS Thyroid Reporting System for Thyroid Nodules. Radiology. 2022 Oct;305(1):149-159. doi: 10.1148/radiol.212319. Epub 2022 Jun 14. PMID 35699576
- [Background] Zhang Y, Zhou P, Tian SM, Zhao YF, Li JL, Li L. Usefulness of combined use of contrast-enhanced ultrasound and TI-RADS classification for the differentiation of benign from malignant lesions of thyroid nodules. Eur Radiol. 2017 Apr;27(4):1527-1536. doi: 10.1007/s00330-016-4508-y. Epub 2016 Aug 15. PMID 27525973